CLINICAL TRIAL: NCT04714671
Title: Effect of Social Stress in the Physiology and Cognition of Suicide Attempters: Heart Rate, Endocrine and Inflammatory Response, Decision Making
Brief Title: Social Stress and Suicide
Acronym: SUPHY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RECHMPL20_0413; 2020-A03045-34 (Other: ANSM)
Record Dates: First submitted 2020-12-21; First posted 2021-01-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Past Major Depressive Episode; Euthymic
Keywords: Suicide; Social stress; Cardiovascular; Decision making; Neuroendocrinology
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Euthymics patients with history of suicide attempt (suicide attempters) (Experimental): Euthymics patients with a lifetime history of suicide attempt will be evaluated using the Structured interview for psychiatric disorder; Columbia-Suicide severity rating scale; Inventory of Depressive Symptoms (IDSC); Young Mania Rating Scale (YMRS).
  Interventions: Other: The virtual version of the Social stress task : V-TSST
- Euthymics patients without any history of suicide attempt (affective controls) (Experimental): Euthymics patients without history of suicide attempt will be evaluated using the Structured interview for psychiatric disorder; Columbia-Suicide severity rating scale; Inventory of Depressive Symptoms (IDSC); Young Mania Rating Scale (YMRS).
  Interventions: Other: The virtual version of the Social stress task : V-TSST

INTERVENTIONS:
Other: The virtual version of the Social stress task : V-TSST — The task consists in a brief presentation about the abilities of participants followed by an arithmetic task in front of a virtual 3D audience projected and one researcher in a small room.First, participants have 5 minutes to prepare an exhibition about their qualities, their strengths and defects, and, why they identify with them. During this period virtual reality shows a closed curtain, and sounds from the audience can be heard. In the second phase, the curtain is raised and the participant must expose his speech during 5 minutes. Audience will remain attentive during 2 minutes, then audience will change to a restless attitude. The third phase consists of subtracting back a two-digit number from a four-digit number, as quickly as possible, starting again if participant makes a mistake. A debriefing of the test is scheduled at the end of the protocol, to remind patients of the purely fictional nature of this test. The visit will only end after a return to the baseline emotional state

SUMMARY:
Only vulnerable patients, when facing environmental stressors, attempt or commit suicide. Previous research demonstrated that suicide attempters usually misunderstand the social context and show impairments in decision making. Heart activity, endocrine and inflammatory response to stress were related with these features. For that, suicide attempters, in a context of social stress, would have maladaptive physiological response impacting the following decision making. The main aim is to identify the physiological response (autonomous nervous system, endocrine and inflammatory response) of suicide attempters under social stress conditions and to investigate the association of this response with the posterior decision making.

The study aims to compare physiological response to social stress and posterior decision-making response in 80 euthymics women with a past mood disorder according to their history of suicide attempt

DETAILED DESCRIPTION:
Hypothesis: 1. suicide attempters will have a lower cortisol, and, greater alpha-amylase and peripheral inflammatory response after a social stressor, compared to non-attempters 2. suicide attempters will have a hyper-activation of the cardiovascular response during the social stressor and a slower recovery to basal levels, compared with non-attempters.

3. With respect to decision-making, suicide attempters will demonstrate riskier decision-making than non-attempters after the social stressor, compared to non-attempters. Risk-taking behavior will be related with lower cortisol and higher testosterone levels after the stressor.

Measures: electrocardiogram (ECG) and impedance cardiography (IKG) will be used to analyse cardiovascular function during social stressor. Salivary samples to analyze cortisol, testosterone and α-amylase. Blood samples to analyze several peripheral inflammatory proteins. The Iowa Gambling Task a neuropsychologial task to evaluate decision making. Several questionnaires of mood, anxiety and psychological pain during the stressor. And a comprehensive battery of clinical measures for screening and assessment of construct of suicide, and psychiatric and social status.

Procedures: Depressed females will be screened and assigned to 2 groups: 1) 40 depressed with suicide attempt history. 2) 40 depressed without suicide attempt history. Participants will confront a virtual version of the Trier Social Stress Test (V-TSST). This test consists in a preparation and execution of a presentation in front of a virtual tribunal for obtain a job position followed by an arithmetic mental task. During the procedure, ECG and IKG will be performed, 5 salivary samples and 5 blood samples (before and after the stressor) and some self-reports of mood, anxiety and pain. After procedure decision making will be assessed. Their participation will consist of 3 visits : inclusion visit (psychiatric interview), visit between 1 to 8 days (social stressor procedure), at 12 months (follow up).

Potential impact and next steps: Identifying differences between the two depressed groups in the physiological response to social stress and their subsequent decision making will advance the understanding of the pathophysiological mechanisms of suicide. As social stress is present in several life events during lifetime, know how suicidal people respond to these issues may help in the implementation of preventive interventions.

ELIGIBILITY:
Inclusion Criteria:

* past major depressive episode according to the DSM-5 criteria (Diagnostic and Statistical Manual of Mental Disorders)
* euthymic (IDSC < 14 and YMRS < 7)
* ability to understand experimental procedures
* able to speak, read and understand French
* able to give written informed consent
* for suicide attempters only: Lifetime history of suicide attempt.
* for affective controls only: No lifetime history of suicide attempt

Exclusion Criteria:

* Lifetime diagnosis of schizoaffective disorder, schizophrenia or social phobia throughout
* Menopause
* Alcohol or illicit substance use disorder in the last 6 months;
* Diagnosis of current cardiovascular (arrhythmia, hypertension, heart valve problems, past heart attack or stroke, congenital heart disease), respiratory (chronic obstructive pulmonary disease, asthma, cystic fibrosis, tuberculosis, lung tumor) endocrine (adrenal disorder, cushing syndrome, adrenal tumor, type-2 diabetes, androgen deficiency, congenital adrenal hyperplasia, hypogonadism, polycystic ovarian syndrome) or neurological disease (dementia, brain stroke, epilepsia, multiple sclerosis, huntington disease, muscular dystrophy, brain or spinal cord tumor, meningitis) based on the first interview, which can interfere with the cardiovascular, endocrine or neurocognitive outcomes of the study;
* current cardiovascular medication which directly affects heart or arterial function or corticoids intake; anticoagulants, antiplatelet agents and dual antiplatelet therapy, angiotensin-converting enzyme inhibitors, angiotensin II receptor blockers, angiotensin-receptor neprilysin inhibitors, beta blockers, calcium channel blockers, vasodilators.
* Pregnancy (urine pregnancy test) or breastfeeding
* refusing to participate
* being in exclusion period for another study
* not being affiliated to the French National Social Security System
* having reached 4500€ annual compensation for participating to clinical trials
* being protected by law or deprived of liberty

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2021-01-27 (Actual); Primary Completion 2025-02-11 (Actual); Study Completion 2025-02-11 (Actual)

PRIMARY OUTCOMES:
Change in salivary cortisol | at visit between 1 to 8 days
  study of the change in salivary cortisol, across all procedure (from -10 to +15, +30, +45 and +60 minutes following the completion of V-TSST)

SECONDARY OUTCOMES:
Changes in cardiovascular response (heart rate) | at visit between 1 to 8 days
  study of the changes in heart rate (HR) from -10 to +15, +30, +45 and +60 minutes following the completion of V-TSST.
Changes in cardiovascular response (Cardiac output) | at visit between 1 to 8 days
  study of the changes in Cardiac output (CO) from -10 to +15, +30, +45 and +60 minutes following the completion of V-TSST.
Changes in cardiovascular response (Total peripheral resistance) | at visit between 1 to 8 days
  study of the changes in Total peripheral resistance (TPR) from -10 to +15, +30, +45 and +60 minutes following the completion of V-TSST.
Changes in cardiovascular response ((time between the two R peaks) | at visit between 1 to 8 days
  study of the changes in R-R interval (time between the two R peaks) from -10 to +15, +30, +45 and +60 minutes following the completion of V-TSST.
Changes in cardiovascular response (pre-ejection period) | at visit between 1 to 8 days
  study of the changes in pre-ejection period (PEP) from -10 to +15, +30, +45 and +60 minutes following the completion of V-TSST.
Changes in cardiovascular response ( Vascular contractibility) | at visit between 1 to 8 days
  study of the changes in Vascular contractibility (VC) from -10 to +15, +30, +45 and +60 minutes following the completion of V-TSST.
Changes in cardiovascular response (High frequency) | at visit between 1 to 8 days
  study of the changes in High frequency (HF) from -10 to +15, +30, +45 and +60 minutes following the completion of V-TSST.
Changes in cardiovascular response (Low frequency) | at visit between 1 to 8 days
  study of the changes in Low frequency (LF) from -10 to +15, +30, +45 and +60 minutes following the completion of V-TSST.
Changes in cardiovascular response (Very low frequency) | at visit between 1 to 8 days
  study of the changes in very Low frequency (VLF) from -10 to +15, +30, +45 and +60 minutes following the completion of V-TSST.
Changes in cardiovascular response (Root mean squared of successive R-R interval differences) | at visit between 1 to 8 days
  study of the changes in Root mean squared of successive R-R interval differences (RMSSD) from -10 to +15, +30, +45 and +60 minutes following the completion of V-TSST.
Changes in salivary testosterone | at visit between 1 to 8 days
  Study of the changes in salivary testosterone, after V-TSST, from -10 to +15, +30, +45 and +60 minutes following the completion fo V-TSST
Changes in salivary α-amylase | at visit between 1 to 8 days
  Study of the changes in salivary α-amylase, after V-TSST, from -10 to +15, +30, +45 and +60 minutes following the completion fo V-TSST
Risk Taking decision making after V-TSST | at visit between 1 to 8 days
  risk-taking using Iowa Gambling (IG) index from Iowa Gambling Task (IGT)
Sense of fairness/unfairness after V-TSST | at visit between 1 to 8 days
  Using the total score of Ultimatum
Domination/submission after V-TSST | at visit between 1 to 8 days
  Using the total score of Hawk and Dove game. The score ranges from 0 to 24, a higher score indicates the most dominant
Changes in anxiety level induced by V-TSST | at visit between 1 to 8 days
  Changes in psychometric state measures : anxiety using the state anxiety inventory, after V-TSST, from -10 to + 15, + 60 and + 120 minutes post V-TSST
Changes in depression level induced by V-TSST | at visit between 1 to 8 days
  Changes in psychometric state measures : mood using the Positive and Negative Affect Schedule, after V-TSST, from baseline to + 15, + 60 and + 120 minutes post V-TSST
Changes in psychological pain level induced by V-TSST | at inclusion
  Changes in psychometric state measures : psychological pain using a visual analogue scale, after V-TSST, from baseline to + 15, + 60 and + 120 post V-TSST. The score ranges from 0 to 10, a higher score indicates the most important psychological pain
Changes in suicidal ideation level induced by V-TSST | at visit between 1 to 8 days
  Changes in psychometric state measures : suicidal ideation using a visual analogue scale, after V-TSST, from baseline to + 15, + 60 and + 120 post V-TSST. SST. The score ranges from 0 to 10, a higher score indicates the most important suicidal ideation
Changes in social distress level induced by V-TSST | at visit between 1 to 8 days
  Changes in psychometric state measures : social distress using a visual analogue scale, after V-TSST, from -10 to + 15, + 60 and + 120 minutes post V-TSST. The score ranges from 0 to 10, a higher score indicates the most important social distress
Changes in C-Reactive Protein (CRP) induced by V-TSST | at visit between 1 to 8 days
  Study of the changes in CRP, after the V-TSST, from -10 to +15, +60, +90 and +120 minutes following the completion post V-TSST.
Changes in Interleukin (IL) - 1b induced by V-TSST | at visit between 1 to 8 days
  Study of the changes in IL-1b, after the V-TSST, from -10 to +15, +60, +90 and +120 minutes following the completion post V-TSST.
Changes in IL-6 induced by V-TSST | at visit between 1 to 8 days
  Study of the changes in IL-6, after the V-TSST, from -10 to +15, +60, +90 and +120 minutes following the completion post V-TSST.
Changes in IL1β induced by V-TSST | at visit between 1 to 8 days
  Study of the changes in IL1β, after the V-TSST, from -10 to +15, +60, +90 and +120 minutes following the completion post V-TSST.
Changes in IL2 induced by V-TSST | at visit between 1 to 8 days
  Study of the changes in IL2, after the V-TSST, from -10 to +15, +60, +90 and +120 minutes following the completion post V-TSST.
Changes in IL4 induced by V-TSST | at visit between 1 to 8 days
  Study of the changes in IL4, after the V-TSST, from -10 to +15, +60, +90 and +120 minutes following the completion post V-TSST.
Changes in IL8 induced by V-TSST | at visit between 1 to 8 days
  Study of the changes in IL8, after the V-TSST, from -10 to +15, +60, +90 and +120 minutes following the completion post V-TSST.
Changes in IL10 induced by V-TSST | at visit between 1 to 8 days
  Study of the changes in IL10, after the V-TSST, from -10 to +15, +60, +90 and +120 minutes following the completion post V-TSST.
Changes in IL13 induced by V-TSST | at visit between 1 to 8 days
  Study of the changes in IL13, after the V-TSST, from -10 to +15, +60, +90 and +120 minutes following the completion post V-TSST.
Changes in IL27 induced by V-TSST | at visit between 1 to 8 days
  Study of the changes in IL27, after the V-TSST, from -10 to +15, +60, +90 and +120 minutes following the completion post V-TSST.
Changes in NF-KB protein induced by V-TSST | at visit between 1 to 8 days
  Study of the changes in NF-KB protein, after the V-TSST, from -10 to +15, +60, +90 and +120 minutes following the completion post V-TSST.
Changes in IKB protein induced by V-TSST | at visit between 1 to 8 days
  Study of the changes in IKB protein, after the V-TSST, from -10 to +15, +60, +90 and +120 minutes following the completion post V-TSST.
Changes in Tumor necrosis factor (TNF) - α protein induced by V-TSST | at visit between 1 to 8 days
  Study of the changes in TNF-α, after the V-TSST, from -10 to +15, +60, +90 and +120 minutes following the completion post V-TSST.
Changes in Interferon (IFN) - γ induced by V-TSST | at visit between 1 to 8 days
  Study of the changes in IFN-γ, after the V-TSST, from -10 to +15, +60, +90 and +120 minutes following the completion post V-TSST.
Changes in Vascular endothelial growth factor (VEGF) induced by V-TSST | at visit between 1 to 8 days
  Study of the changes in VEGF, after the V-TSST, from -10 to +15, +60, +90 and +120 minutes following the completion post V-TSST.
Changes in kyrunenine induced by V-TSST | at visit between 1 to 8 days
  Study of the changes in kyrunenine, after the V-TSST, from -10 to +15, +60, +90 and +120 minutes following the completion post V-TSST.
Changes in sCD62P induced by V-TSST | at visit between 1 to 8 days
  Study of the changes in sCD62P, after the V-TSST, from -10 to +15, +60, +90 and +120 minutes following the completion post V-TSST.
Changes in sCD40L induced by V-TSST | at visit between 1 to 8 days
  Study of the changes in sCD40L, after the V-TSST, from -10 to +15, +60, +90 and +120 minutes following the completion post V-TSST.
Changes in Platelet factor (PF) 4 induced by V-TSST | at visit between 1 to 8 days
  Study of the changes in PF4, after the V-TSST, from -10 to +15, +60, +90 and +120 minutes following the completion post V-TSST.
Changes in RANTES induced by V-TSST | at visit between 1 to 8 days
  Study of the changes in RANTES, after the V-TSST, from -10 to +15, +60, +90 and +120 minutes following the completion post V-TSST.
Changes in Brain derived neurotrophic factor (BDNF) induced by V-TSST | at visit between 1 to 8 days
  Study of the changes in BDNF, after the V-TSST, from -10 to +15, +60, +90 and +120 minutes following the completion post V-TSST.
Changes in sOx40L induced by V-TSST | at visit between 1 to 8 days
  Study of the changes in sOx40L, after the V-TSST, from -10 to +15, +60, +90 and +120 minutes following the completion post V-TSST.
Changes in Microparticle induced by V-TSST | at visit between 1 to 8 days
  Study of the changes in Microparticle, after the V-TSST, from -10 to +15, +60, +90 and +120 minutes following the completion post V-TSST.
Changes in Mitochondrial deoxyribonucleic acid (DNA) of platelet origin induced by V-TSST | at visit between 1 to 8 days
  Study of the changes in Mitochondrial DNA of platelet origin, after the V-TSST, from -10 to +15, +60, +90 and +120 minutes following the completion post V-TSST.
Suicidal behavior evaluated with the C-SSRS | at 12 months post V-SST

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Montpellier, Montpellier, Hérault, France